CLINICAL TRIAL: NCT06265415
Title: A Comparative Study of Intravenous Labetalol Versus Intravenous Nitroglycerin Versus Sublingual Nifedipine to Control Blood Pressure in Severe Pre-eclampsia
Brief Title: Comparative Study of Intravenous Labetalol Versus Intravenous Nitroglycerin Versus Sublingual Nifedipine
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Diaa Aly Abdelaal, Resident-anesthesia,surgical intensive care and pain control department-sohag hospital university, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-01-07MS
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Severe Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — Labetalol; Nitroglycerin; Nifedipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group A (Active Comparator): (20 patients) will receive Labetalol intravenous infusion. The starting infusion rate is 5mg/h,the infusion rate will be changed 1mg/h up every 10 minutes until the desired goal achieved which is a decrease in systolic blood pressure (SBP) to 120 - 140 mmHg and a decrease in diastolic blood pressure (DBP) to 80 - 90 mmHg every 10 minutes
  Interventions: Drug: Labetalol
- group B (Active Comparator): (20 patients) will receive calculated dose of Nitroglycerine started as intravenous infusion, The starting infusion rate is 4.8mg/h ,the infusion rate will be changed 1mg/h every 10 minutes up until the therapeutic goal achieved, which is a decrease in systolic blood pressure (SBP) to 120 - 140 mmHg and a decrease in diastolic blood pressure (DBP) to 80 - 90 mmHg
  Interventions: Drug: Nitroglycerine
- group C (Active Comparator): , (20 patients) will receive calculated dose of nifedipine the content (100 µL) of a 10 mg capsule of nifedipine was drawn up into an insulin syringe and deposited sublingually, every 30 min.( Maximum dose of nifedipine 120 mg/day) ) until the therapeutic goal achieved, which is a decrease in systolic blood pressure (SBP) to 120 - 140 mmHg and a decrease in diastolic blood pressure (DBP) to 80 - 90 mmHg
  Interventions: Drug: Nifedipine

INTERVENTIONS:
Drug: Labetalol — it contains both selective, competitive, alpha1-adrenergic antagonism and non-selective, competitive, beta-adrenergic (B1 and B2) blocking activity in a single agent
  Arms: group A
Drug: Nitroglycerine — a nitric oxide donor with low oral bioavailability and a very short half-life, has a potent venodilator effect in low doses and affects arterial tone at high doses
  Arms: group B
Drug: Nifedipine — dihydropyridine calcium channel blocker. Its main uses are as an antianginal and antihypertensive
  Arms: group C

SUMMARY:
Pre-eclampsia (PE) is one of the most frequent pregnancy complications and is one of the main causes of maternal and fetal morbidity and mortality in its severe form.control of blood pressure is of crucial importance to avoid maternal and fetal complications.Therapeutic modalities that can target the underlying pathophysiological changes and reverse the endothelial dysfunction could help to ameliorate the systemic manifestations in patients with severe PE. Either Intravenous labetalol and nitroglycerine as well as sublingual nifedipine have been frequantly used for the management of acute severe hypertension in PE

DETAILED DESCRIPTION:
Pre-eclampsia (PE) is one of the most frequent pregnancy complications and is one of the main causes of maternal and fetal morbidity and mortality in its severe form.

Pre-eclampsia characterized by

* Rising blood pressure (BP ≥ 140/90 that occurs after 20 weeks of gestation in a woman with previously normal BP.
* . Proteinuria (≥300mg/24hr . This correlates with 30mg/dl or ≥1+ on urine dipstick)
* Edema control of blood pressure is of crucial importance to avoid maternal and fetal complications.

The pathophysiology of pre-eclampsia is most likely inadequate placentation, leading to endothelial dysfunction and reduced nitric oxide bioavailability. Therapeutic modalities that can target the underlying pathophysiological changes and reverse the endothelial dysfunction could help to ameliorate the systemic manifestations in patients with severe PE. Either Intravenous labetalol and nitroglycerine as well as sublingual nifedipine have been frequantly used for the management of acute severe hypertension in PE

. Nitroglycerine, a nitric oxide donor with low oral bioavailability and a very short half-life, has a potent venodilator effect in low doses and affects arterial tone at high doses Labetalol is useful as it contains both selective, competitive, alpha1-adrenergic antagonism and non-selective, competitive, beta-adrenergic (B1 and B2) blocking activity in a single agent Nifedipine is a dihydropyridine calcium channel blocker. Its main uses are as an antianginal and antihypertensive

ELIGIBILITY:
Inclusion Criteria:

* The study will include 60 adult female patients ( 18 to 40 years old) with sever pre-eclampsia, who were being managed with MgSO4 loading and maintenance doses Severe hypertension was diagnosed by Systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥110 mmHg.

Mean arterial blood pressure ≥ 127 mmHg

Exclusion Criteria:

1. Patient refusal.
2. Eclampsia
3. Emenant eclampsia
4. HELLP syndrome
5. Chronic hypertension
6. Patients who have chronic obstructive pulmonary disease.
7. Patient with acute or chronic liver failure.
8. Known allergy to the study medications

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
duration of control blood pressure | 1 year
  duration required, of nitroglycerin compared to labetalol and sublingual nifedipine in terms of acute control of blood pressure in severe PE.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Mulhim AA, Abu-Heija A, Al-Jamma F, El-Harith el-HA. Pre-eclampsia: maternal risk factors and perinatal outcome. Fetal Diagn Ther. 2003 Jul-Aug;18(4):275-80. doi: 10.1159/000070809. PMID 12835589
- [Background] Olayinka L, Garnett E, Burnett B, Devaraj S. Comparison of random urine protein/creatinine ratio with 24-hour urine protein in suspected pre-eclampsia. Pract Lab Med. 2023 Jun 21;36:e00316. doi: 10.1016/j.plabm.2023.e00316. eCollection 2023 Aug. PMID 37649542
- [Background] Johal T, Lees CC, Everett TR, Wilkinson IB. The nitric oxide pathway and possible therapeutic options in pre-eclampsia. Br J Clin Pharmacol. 2014 Aug;78(2):244-57. doi: 10.1111/bcp.12301. PMID 24313856
- [Background] Divakaran S, Loscalzo J. The Role of Nitroglycerin and Other Nitrogen Oxides in Cardiovascular Therapeutics. J Am Coll Cardiol. 2017 Nov 7;70(19):2393-2410. doi: 10.1016/j.jacc.2017.09.1064. PMID 29096811